CLINICAL TRIAL: NCT00655447
Title: Ovarian Conservation: Long-Term Health Outcomes From the Nurse's Health Study.
Brief Title: Examining the Long-Term Risks of Oophorectomy
Status: Completed | Type: Observational
Sponsor: Parker, William H., M.D. (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: William Parker, John Wayne Cancer Institute
Other Study IDs: PARW-OVCONS-0307
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Heart Disease; Stroke; Breast Cancer; Ovarian Cancer; Cancer; Hip Fracture; Death
Keywords: oophorectomy; ovarian conservation; stroke; breast cancer; ovarian cancer; other cancer; hip fracture
MeSH Terms: conditions — Coronary Disease; Stroke; Breast Neoplasms; Ovarian Neoplasms; Neoplasms; Hip Fractures; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: all women having a hysterectomy with oophorectomy
- 2: all women having a hysterectomy without removal of ovaries

SUMMARY:
At the time of hysterectomy for benign disease, the overall health benefits of preserving ovarian function in a large population of women have not been established.

DETAILED DESCRIPTION:
We are conducting a prospective, observational study of 32,175 women participants of the Nurse's Health Study who had a hysterectomy with or without removal of both ovaries. We are evaluating mortality and morbidity due to the following conditions: coronary heart disease, stroke, breast cancer, ovarian cancer, other cancer, hip fracture and death from all causes.

ELIGIBILITY:
Inclusion Criteria:

* Women who had hysterectomies were classified into simple hysterectomy or hysterectomy with both ovaries removed.

Exclusion Criteria:

* Evidence of cancer, coronary heart disease (MI or Angina Pectoris), stroke, or hip fracture before entering the study were excluded. Cancer as an indication for hysterectomy also excluded.
* Women reporting unilateral oophorectomy, unknown oophorectomy status, unknown age of hysterectomy, or those who had oophorectomy before hysterectomy were excluded.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nurses' Health Study I, which included 122,701 married registered nurses living in 11 U.S. states and who were ages 30 to 55 in 1976
Sampling Method: Non-Probability Sample
Enrollment: 32175 (Actual)
Dates: Start 1980-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
mortality and morbidity due to the following conditions: coronary heart disease, stroke, breast cancer, ovarian cancer, other cancer, hip fracture and death from all causes. | 28 years

SECONDARY OUTCOMES:
The effect of postmenopausal hormone use on mortality and morbidity due to the following conditions: coronary heart disease, stroke, breast cancer, ovarian cancer, other cancer, hip fracture and death from all causes. | 28 years

CONTACTS AND LOCATIONS:
Overall Officials: William H Parker, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Parker, Rosenman, Rodi Gynecology Group, Santa Monica, California, United States

REFERENCES:
- [Background] Parker WH, Broder MS, Liu Z, Shoupe D, Farquhar C, Berek JS. Ovarian conservation at the time of hysterectomy for benign disease. Obstet Gynecol. 2005 Aug;106(2):219-26. doi: 10.1097/01.AOG.0000167394.38215.56. PMID 16055568